CLINICAL TRIAL: NCT04291196
Title: Virtual Reality as a Tool to Reduce Pre-procedure Anxiety Prior ECT Via Enhancing Patient Education
Brief Title: Virtual Reality to Reduce Pre-procedure Anxiety Prior ECT
Acronym: PERFECT-VR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 036-2019
Record Dates: First submitted 2019-11-12; First posted 2020-03-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: ECT; Electroconvulsive Therapy; Virtual Reality; Anxiety; Education; Hemodynamics; Depression; Cognition; Mental Health
MeSH Terms: conditions — Anxiety Disorders; Depression; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive Virtual Reality (Experimental): Patients will be immersed in the ECT experience using VR-ECT 360o video (VR-ECT).
  Interventions: Other: VR-ECT 360o Video
- Standard Treatment (Other): Patients will receive standard preparation for their ECT session.
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Other: VR-ECT 360o Video — Patients in the VR arm will be immersed in the ECT process in first person utilizing Google Cardboard headsets. Patients will experience in 360 entering the procedure room, IV insertion, pretreatment checks, anesthetic induction followed by induction of seizure, and recovery. The experience will also have voice-over narration simultaneously describing the procedure and its risks and benefits.
  Arms: Immersive Virtual Reality
Other: Standard Treatment — Patients will receive preparation for their ECT as per standard of care, i.e. a discussion with a Psychiatrist.
  Arms: Standard Treatment

SUMMARY:
Lack of patient knowledge about ECT (electroconvulsive therapy) is a leading cause of treatment fear with 60% of ECT patients reporting high levels of anxiety.

The purpose of this study is to determine if using Virtual Reality (VR) to allow patients' to experience a virtual ECT education session before treatment is useful in lowering treatment anxiety and increasing knowledge about ECT if compared to standard treatment. In addition, measuring heart rate and blood pressure levels before ECT treatment will allow us to assess changes in anxiety levels.

Individuals who choose to participate will be placed (participant will have a 50% chance to be placed in either group) to view either a virtual reality video to experience a virtual ECT session, or to receive standard preparation, i.e. a discussion with a psychiatrist. Before and after this session participants will be asked to complete a measurement of their anxiety level and knowledge about ECT (ECT Attitude & Knowledge Questionnaire). Just before ECT treatment, blood pressure, heart rate and anxiety level will be measured. Participants will also complete cognitive and depression assessments.

This study will help to develop a relationship between healthcare providers and patients and their families to help with education before ECT treatment.

DETAILED DESCRIPTION:
Virtual reality (VR) is increasingly being used in healthcare, in particular as a form of exposure therapy for patients with psychiatric disorders. It immerses patients into hospital-based procedures. We and others showed that VR prep reduces anxiety levels for elective surgical patients (manuscript submitted). However, the efficacy of VR in reducing peri-procedural anxiety in vulnerable psychiatric populations has not been assessed. This will be the first RCT utilizing VR to reduce patient anxiety before ECT through education. If VR education reduces anxiety in this vulnerable population (as proof of concept), it could increase ECT success by decreasing anesthetic requirements. Using VR technology, our study will provide patients and their families with a balanced and in-depth look at ECT safety and efficacy, and its recent advances in management of psychiatric disorders.

Primary objectives of this study are to assess whether creating a VR-ECT-360 video that immerses and educates patients and their families in the ECT experience 1) enhances factual knowledge and reduces stigmatizing attitudes toward ECT, and 2) reduces pre-procedure anxiety as compared to traditional 2D video. The secondary objective is to investigate the ease of use of VR technology in a vulnerable psychiatric patient population. Given the high rate of treatment refusals in this population, we hypothesize that implementation of our approach will reduce anxiety through patient education thereby decreasing chances for treatment refusal and drop-out rates. We suggest that use of VR will be a clinically relevant approach in such a vulnerable population (as proof of concept) and could increase ECT success by decreasing anesthetic requirements (anesthetics suppress desired seizure activity).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* First time undergoing ECT within the last year
* Outpatient/inpatient recommended for ECT
* Within 2-4 days of ECT procedure or no ECT within the past year
* Referred by psychiatrist
* Able to understand English
* Able to watch and respond to questions

Exclusion Criteria:

* Lack of patient consent or capacity to give consent
* Visual and hearing impairments precluding the ability to watch or listen to video
* History of significant motion sickness (i.e. occur during exposure to physical, visual and virtual motion, cybersickness verbally declared by patient)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Pre-operative Anxiety | Measurement completed 1) up to 2-3 days before ECT education 2) right after ECT education 3) prior to ECT (day of proceudre)
  Change in pre-operative anxiety will be assessed using the Visual Anxiety Scale (VAS, Not at all anxious to extremely anxious).
Change in ECT Knowledge | Measurement completed 1) Immediately Before ECT education 2) Immediately After ECT education 3) Immediately Prior to ECT
  Change in ECT knowledge will be assessed using the ECT Attitude & Knowledge Questionnaire.
Heart rate | Measurement completed prior to ECT session on the day of procedure.
  Heart rate will be measured in beats/min
Mean arterial blood pressure | Measurement completed prior to ECT session on the day of procedure.
  Mean arterial blood pressure will be measured in mmHg.

SECONDARY OUTCOMES:
Cognitive Performance | Measurement completed 1) Before intervention on the day of procedure 2) Prior to ECT on the day of procedure
  Cognitive performance will be assessed using the Montreal Cognitive Assessment (MoCA).
Depression | Measurement completed 1) Before intervention on the day of procedure 2) Prior to ECT on the day of procedure
  Depression will be assessed.
Ease of Use of VR Technology | Measurement completed immediately after ECT education on the day of procedure.
  Ease of use of VR technology will be assessed using the system usability, scale (SUS), only in VR arm.

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Alam, Principal Investigator — SHSC
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No